CLINICAL TRIAL: NCT02614261
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study of LY2951742 in Patients With Chronic Migraine - the REGAIN Study
Brief Title: Evaluation of Galcanezumab in the Prevention of Chronic Migraine
Acronym: REGAIN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15769; I5Q-MC-CGAI (Other: Eli Lillly and Company); 2015-001883-21 (EudraCT Number)
Record Dates: First submitted 2015-11-23; First posted 2015-11-25 (Estimated); Results first posted 2019-01-07 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-04

CONDITIONS: Chronic Migraine
Keywords: prevention; prophylaxis; headache
MeSH Terms: conditions — Headache | interventions — galcanezumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (Placebo Comparator): * Double-blind treatment phase: Participants received placebo once a month by subcutaneous (SC) injection for 3 months.
  * Open-label extension phase: After completion of double-blind phase, participants had an option to enter open-label extension phase where they receive 240 milligram (mg) galcanezumab SC at first month, 120mg at second month followed by 120mg or 240mg once a month (at the discretion of the investigator) for the remaining 7 months.
  * Follow-up phase: After completion or discontinuation from double-blind or open-label extension phases, participants entered follow-up phase where they were observed for 4 months. No treatments administered.
  Interventions: Drug: Galcanezumab; Drug: Placebo
- Galcanezumab 120 mg (Experimental): * Double-blind treatment phase: Participants received loading dose of 240 mg of galcanezumab at first dosing visit followed 120 mg galcanezumab once a month by SC injection for 2 months.
  * Open-label extension phase: After completion of double-blind phase, participants had an option to enter open-label extension phase where they received 240mg galcanezumab SC at first month, 120mg at second month followed by 120mg or 240mg once a month (at the discretion of the investigator) for the remaining 7 months.
  * Follow-up phase: After completion or discontinuation from double-blind or open-label extension phases, participants entered follow-up phase where they were observed for 4 months. No treatments administered.
  Interventions: Drug: Galcanezumab
- Galcanezumab 240 mg (Experimental): * Double-blind treatment phase: Participants received 240 mg of galcanezumab once a month by subcutaneous injection for 3 months.
  * Open-label extension phase: After completion of double-blind phase, participants had an option to enter open-label extension phase where they received 240mg galcanezumab SC at first month, 120mg at second month followed by 120mg or 240mg once a month (at the discretion of the investigator) for the remaining 7 months.
  * Follow-up phase: After completion or discontinuation from double-blind or open-label extension phases, participants entered follow-up phase where they were observed for 4 months. No treatments administered.
  Interventions: Drug: Galcanezumab
- Israel Addendum (Experimental): Eligible participants from main study were enrolled in Israel addendum. Participants received 120mg or 240mg galcanezumab SC once a month, at the discretion of the investigator, for up to 3 years or until Israel's Ministry of Health's conditions for continued access cease to be met, whichever occurs first.
  Interventions: Drug: Galcanezumab

INTERVENTIONS:
Drug: Galcanezumab — Administered SC
  Other Names: LY2951742
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
The main purpose of this study is to evaluate the efficacy of the study drug known as galcanezumab in participants with chronic migraine.

ELIGIBILITY:
Inclusion Criteria:

Main Study:

* Have a diagnosis of chronic migraine as defined by International Headache Society (IHS) International Classification of Headache Disorders (ICHD)-3 beta guidelines (1.3) (ICHD-3 2013), with a history of migraine headaches of at least 1 year prior to screening, and migraine onset prior to age 50.

Israel addendum:

* Participants must have completed all phases of main study, including the 4-month post-treatment follow-up phase, during which no investigational product was administered.
* Participants also must be considered by the investigator to have benefited from galcanezumab treatment and must have exhausted alternative therapies for the prevention of migraine.

Exclusion Criteria:

* Are currently enrolled in or have participated within the last 30 days or within 5 half-lives (whichever is longer) in a clinical trial involving an investigational product.
* Current use or prior exposure to galcanezumab or another calcitonin gene-related peptide (CGRP) antibody.
* Known hypersensitivity to multiple drugs, monoclonal antibodies or other therapeutic proteins, or to galcanezumab.
* History of persistent daily headache, cluster headache or migraine subtypes including hemiplegic (sporadic or familial) migraine, ophthalmoplegic migraine, and migraine with brainstem aura (basilar-type migraine) defined by IHS ICHD-3 beta.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1117 (Actual)
Dates: Start 2015-11-30 (Actual); Primary Completion 2017-03-16 (Actual); Study Completion 2021-07-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (103):
- United States (52):
  - 21st Century Neurology, Phoenix, Arizona
  - Arizona Research Center, Phoenix, Arizona
  - Pharmacology Research Institute, Encino, Encino, California
  - Fullerton Neurology and Headache Center, Fullerton, California
  - Pharmacology Research Institute, Los Alamitos, Los Alamitos, California
  - Pharmacology Research Institute, Newport Beach, Newport Beach, California
  - Desert Valley Research, Rancho Mirage, California
  - Anderson Clinical Research, Redlands, California
  - Artemis Institute for Clinical Research, San Diego, California
  - Medical Center for Clinical Research, San Diego, California
  - Optimus Medical Group, San Francisco, California
  - Colorado Neurological Institute, Englewood, Colorado
  - Advanced Neurosciences Research, LLC, Fort Collins, Colorado
  - Associated Neurologists of Southern Connecticut, Fairfield, Connecticut
  - Avail Clinical Research LLC, DeLand, Florida
  - Clinical Neuroscience Solutions Inc, Jacksonville, Florida
  - |Renstar Medical Research, Ocala, Florida
  - Psychiatric Inst of Florida-Clinical Neuroscience Solutions, Orlando, Florida
  - Compass Research, Oviedo, Florida
  - Premiere Research Institute at Palm Beach Neurology, West Palm Beach, Florida
  - Northwest Clinical Trials, Boise, Idaho
  - Christie Clinic, LLC, Champaign, Illinois
  - Robbins Headache Clinic, Riverwoods, Illinois
  - Midwest Institute for Clinical Research, Indianapolis, Indiana
  - Phoenix Medical Research, Inc, Prairie Village, Kansas
  - Heartland Research Associates, Wichita, Kansas
  - PharmaSite Research Inc, Baltimore, Maryland
  - Boston Clinical Trials Inc, Boston, Massachusetts
  - Michigan Head, Pain and Neurological Institute, Ann Arbor, Michigan
  - Clinical Research Institute, Minneapolis, Minnesota
  - Healthcare Research Network - Hazelwood, Hazelwood, Missouri
  - ClinVest, Springfield, Missouri
  - Albuquerque Clinical Trials, Albuquerque, New Mexico
  - Dent Neurological Institute, Amherst, New York
  - Island Neuro Associates,PC, Plainview, New York
  - Univ of Cincinnati College of Medicine, Cincinnati, Ohio
  - Healthcare Research Consultant, Tulsa, Oklahoma
  - Preferred Primary Care Physicians, Pleasant Hills, Pennsylvania
  - Abington Neurological Associates, Willow Grove, Pennsylvania
  - Clinical Trials of South Carolina, Charleston, South Carolina
  - University of South Carolina, Columbia, South Carolina
  - Coastal Carolina Research Center, Inc., Mt. Pleasant, South Carolina
  - BG Neurology, Spartanburg, South Carolina
  - ClinSearch, Chattanooga, Tennessee
  - FutureSearch Trials of Neurology and Sleep Lab, Austin, Texas
  - Headache Medicine Specialist of North Texas, Dallas, Texas
  - Foothill Family Clinic, Salt Lake City, Utah
  - Health Research of Hampton Roads Inc, Newport News, Virginia
  - Sentara Neurology Specialists, Virginia Beach, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington
  - Premier Clinical Research, Spokane, Washington
  - Dean Foundation for Health Research and Education, Middleton, Wisconsin
- Argentina (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Buenos Aires
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ciudad Autonoma de Buenos Aire
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Córdoba
- Canada (4):
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Brampton
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Kelowna
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Montreal
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Ottawa
- Czechia (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brno
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kladno
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Prague
- Germany (9):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Berlin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bielefeld
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bochum
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Essen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kassel
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Königstein
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Prien am Chiemsee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tübingen
- Israel (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hadera
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kfar Saba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ramat Gan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tel Aviv
- Italy (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bologna
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Florence
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Modena
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pavia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Roma
- Mexico (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aguascalientes
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Culiacán
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., México
- Netherlands (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Amsterdam
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leiden
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nijmegen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zwolle
- Puerto Rico (4):
  - Office of Dr. Ruddy Guerra, Manatí
  - GCM Medical Group PSC, San Juan
  - Instituto de Neurologia Dra. Ivonne Fraga, San Juan
  - Neuro GI Wellness Center, San Juan
- Spain (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pamplona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santander
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Valencia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Valladolid
- Taiwan (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kaohsiung City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tainan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taipei
- United Kingdom (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Glasgow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hull
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., London
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Stoke-on-Trent

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Diener HC, Day KA, Lipsius S, Aurora SK, Hindiyeh NA, Detke HC. Shift from chronic to episodic migraine frequency in a long-term phase 3 study of galcanezumab. J Headache Pain. 2025 Feb 3;26(1):26. doi: 10.1186/s10194-025-01956-x. PMID 39901101
- [Derived] Pozo-Rosich P, Detke HC, Wang S, Dolezil D, Li LQ, Aurora SK, Reuter U. Long-term treatment with galcanezumab in patients with chronic migraine: results from the open-label extension of the REGAIN study. Curr Med Res Opin. 2022 May;38(5):731-742. doi: 10.1080/03007995.2022.2059975. Epub 2022 Apr 15. PMID 35392739
- [Derived] Ailani J, Kuruppu DK, Rettiganti M, Oakes T, Schroeder K, Wietecha L, Port M, Blumenfeld AM. Does "wearing off" of efficacy occur in galcanezumab-treated patients at the end of the monthly treatment cycle? Post hoc analyses of four phase III randomized trials. Headache. 2022 Feb;62(2):198-207. doi: 10.1111/head.14257. Epub 2022 Jan 25. PMID 35076090
- [Derived] Citrome L, Sanchez Del Rio M, Dong Y, Nichols RM, Tockhorn-Heidenreich A, Foster SA, Stauffer VL. Benefit-Risk Assessment of Galcanezumab Versus Placebo for the Treatment of Episodic and Chronic Migraine Using the Metrics of Number Needed to Treat and Number Needed to Harm. Adv Ther. 2021 Aug;38(8):4442-4460. doi: 10.1007/s12325-021-01848-x. Epub 2021 Jul 15. PMID 34264500
- [Derived] Pozo-Rosich P, Samaan KH, Schwedt TJ, Nicholson RA, Rettiganti M, Pearlman EM. Galcanezumab Provides Consistent Efficacy Throughout the Dosing Interval Among Patients with Episodic and Chronic Migraine: A Post Hoc Analysis. Adv Ther. 2021 Jun;38(6):3154-3165. doi: 10.1007/s12325-021-01708-8. Epub 2021 May 5. PMID 33950375
- [Derived] Ament M, Day K, Stauffer VL, Skljarevski V, Rettiganti M, Pearlman E, Aurora SK. Effect of galcanezumab on severity and symptoms of migraine in phase 3 trials in patients with episodic or chronic migraine. J Headache Pain. 2021 Feb 6;22(1):6. doi: 10.1186/s10194-021-01215-9. PMID 33549036
- [Derived] Kuruppu DK, North JM, Kovacik AJ, Dong Y, Pearlman EM, Hutchinson SL. Onset, Maintenance, and Cessation of Effect of Galcanezumab for Prevention of Migraine: A Narrative Review of Three Randomized Placebo-Controlled Trials. Adv Ther. 2021 Mar;38(3):1614-1626. doi: 10.1007/s12325-021-01632-x. Epub 2021 Feb 5. PMID 33544305
- [Derived] Dodick DW, Doty EG, Aurora SK, Ruff DD, Stauffer VL, Jedynak J, Dong Y, Pearlman EM. Medication overuse in a subgroup analysis of phase 3 placebo-controlled studies of galcanezumab in the prevention of episodic and chronic migraine. Cephalalgia. 2021 Mar;41(3):340-352. doi: 10.1177/0333102420966658. Epub 2020 Nov 3. PMID 33143451
- [Derived] Ailani J, Andrews JS, Rettiganti M, Nicholson RA. Impact of galcanezumab on total pain burden: findings from phase 3 randomized, double-blind, placebo-controlled studies in patients with episodic or chronic migraine (EVOLVE-1, EVOLVE-2, and REGAIN trials). J Headache Pain. 2020 Oct 17;21(1):123. doi: 10.1186/s10194-020-01190-7. PMID 33069214
- [Derived] Ford J, Tassorelli C, Leroux E, Wang S, Ayer D, Nichols R, Detke H. Changes in patient functioning and disability: results from a phase 3, double-blind, randomized, placebo-controlled clinical trial evaluating galcanezumab for chronic migraine prevention (REGAIN). Qual Life Res. 2021 Jan;30(1):105-115. doi: 10.1007/s11136-020-02623-1. Epub 2020 Sep 15. PMID 32930994
- [Derived] Stauffer VL, Turner I, Kemmer P, Kielbasa W, Day K, Port M, Quinlan T, Camporeale A. Effect of age on pharmacokinetics, efficacy, and safety of galcanezumab treatment in adult patients with migraine: results from six phase 2 and phase 3 randomized clinical trials. J Headache Pain. 2020 Jun 23;21(1):79. doi: 10.1186/s10194-020-01148-9. PMID 32576229
- [Derived] Bangs ME, Kudrow D, Wang S, Oakes TM, Terwindt GM, Magis D, Yunes-Medina L, Stauffer VL. Safety and tolerability of monthly galcanezumab injections in patients with migraine: integrated results from migraine clinical studies. BMC Neurol. 2020 Jan 17;20(1):25. doi: 10.1186/s12883-020-1609-7. PMID 31952501
- [Derived] Kielbasa W, Quinlan T. Population Pharmacokinetics of Galcanezumab, an Anti-CGRP Antibody, Following Subcutaneous Dosing to Healthy Individuals and Patients With Migraine. J Clin Pharmacol. 2020 Feb;60(2):229-239. doi: 10.1002/jcph.1511. Epub 2019 Sep 4. PMID 31482569
- [Derived] Ruff DD, Ford JH, Tockhorn-Heidenreich A, Sexson M, Govindan S, Pearlman EM, Wang SJ, Khan A, Aurora SK. Efficacy of galcanezumab in patients with chronic migraine and a history of preventive treatment failure. Cephalalgia. 2019 Jul;39(8):931-944. doi: 10.1177/0333102419847957. Epub 2019 May 19. PMID 31104507
- [Derived] Forderreuther S, Zhang Q, Stauffer VL, Aurora SK, Lainez MJA. Preventive effects of galcanezumab in adult patients with episodic or chronic migraine are persistent: data from the phase 3, randomized, double-blind, placebo-controlled EVOLVE-1, EVOLVE-2, and REGAIN studies. J Headache Pain. 2018 Dec 29;19(1):121. doi: 10.1186/s10194-018-0951-2. PMID 30594122
- [Derived] Nichols R, Doty E, Sacco S, Ruff D, Pearlman E, Aurora SK. Analysis of Initial Nonresponders to Galcanezumab in Patients With Episodic or Chronic Migraine: Results From the EVOLVE-1, EVOLVE-2, and REGAIN Randomized, Double-Blind, Placebo-Controlled Studies. Headache. 2019 Feb;59(2):192-204. doi: 10.1111/head.13443. Epub 2018 Nov 21. PMID 30462830
- [Derived] Detke HC, Goadsby PJ, Wang S, Friedman DI, Selzler KJ, Aurora SK. Galcanezumab in chronic migraine: The randomized, double-blind, placebo-controlled REGAIN study. Neurology. 2018 Dec 11;91(24):e2211-e2221. doi: 10.1212/WNL.0000000000006640. Epub 2018 Nov 16. PMID 30446596
- See also: A Study of LY2951742 in the Prevention of Chronic Migraine (REGAIN) — https://trials.lillytrialguide.com/en-US/trial/FnCyu97viesEckigw4wmc

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1. Main study: This randomised part of study was conducted in 3 phases
     * a 3-month double-blind treatment phase
     * an optional 9-month open-label extension phase
     * a 4-month follow-up phase
  2. Israel addendum: Participants in Israel who completed all phases in main study, benefited from galcanezumab and had no other suitable alternative treatment options available were provided continued-access to galcanezumab where safety was monitored.
Groups:
- Galcanezumab 120mg: * Double-blind treatment phase: Participants received loading dose of 240 mg of galcanezumab at first dosing visit followed 120 mg galcanezumab once a month by subcutaneous injection for 2 months.
  * Open-label extension phase: After completion of double-blind phase, participants had an option to enter open-label extension phase where they received 240mg galcanezumab SC at first month, 120mg at second month followed by 120mg or 240mg once a month (at the discretion of the investigator) for the remaining 7 months.
  * Follow-up phase: After completion or discontinuation from double-blind or open-label extension phases, participants entered follow-up phase where they were observed for 4 months. No treatments administered.
- Galcanezumab 240mg: * Double-blind treatment phase: Participants received 240 mg of galcanezumab once a month by subcutaneous injection for 3 months.
  * Open-label extension phase: After completion of double-blind phase, participants had an option to enter open-label extension phase where they received 240mg galcanezumab SC at first month, 120mg at second month followed by 120mg or 240mg once a month (at the discretion of the investigator) for the remaining 7 months.
  * Follow-up phase: After completion or discontinuation from double-blind or open-label extension phases, participants entered follow-up phase where they were observed for 4 months. No treatments administered.
Period: Double-Blind Treatment Phase
Arm/Group | Placebo | Galcanezumab 120mg | Galcanezumab 240mg | Israel Addendum
Started | 559 | 279 | 279 | 0
Received at Least One Dose of Study Drug | 558 | 278 | 277 | 0
Safety Population | 558 | 273 (5 participants discontinued after receiving loading dose of 240mg. They were included under 240mg arm for safety analysis.) | 282 | 0
Completed | 509 | 262 | 266 | 0
Not Completed | 50 | 17 | 13 | 0
Not completed — Adverse Event | 7 | 3 | 2 | 0
Not completed — Lack of Efficacy | 4 | 0 | 0 | 0
Not completed — Lost to Follow-up | 9 | 4 | 1 | 0
Not completed — Physician Decision | 2 | 1 | 1 | 0
Not completed — Pregnancy | 2 | 2 | 0 | 0
Not completed — Protocol Violation | 6 | 1 | 0 | 0
Not completed — Screen failure | 0 | 1 | 2 | 0
Not completed — Withdrawal by Subject | 20 | 5 | 7 | 0
Period: Open-Label Extension Phase
Arm/Group | Placebo | Galcanezumab 120mg | Galcanezumab 240mg | Israel Addendum
Started | 501 (Participants from double-blind treatment phase had the option to enter the open-label extension phase or proceed directly to the follow-up phase.) | 259 (Participants from double-blind treatment phase had the option to enter the open-label extension phase or proceed directly to the follow-up phase.) | 262 (Participants from double-blind treatment phase had the option to enter the open-label extension phase or proceed directly to the follow-up phase.) | 0
Safety Population | 501 | 259 | 262 | 0
Completed | 413 | 204 | 208 | 0
Not Completed | 88 | 55 | 54 | 0
Not completed — Adverse Event | 23 | 12 | 11 | 0
Not completed — Lack of Efficacy | 14 | 12 | 14 | 0
Not completed — Lost to Follow-up | 15 | 7 | 9 | 0
Not completed — Physician Decision | 2 | 0 | 0 | 0
Not completed — Pregnancy | 1 | 2 | 1 | 0
Not completed — Protocol Violation | 3 | 4 | 1 | 0
Not completed — Withdrawal by Subject | 30 | 18 | 18 | 0
Period: Follow-up Phase
Arm/Group | Placebo | Galcanezumab 120mg | Galcanezumab 240mg | Israel Addendum
Started | 453 (Participants from double-blind treatment or open-label extension phases entered the follow-up phase.) | 228 (Participants from double-blind treatment or open-label extension phases entered the follow-up phase.) | 231 (Participants from double-blind treatment or open-label extension phases entered the follow-up phase.) | 0
Entered From Double-blind Treatment Phase | 15 | 5 (1 among these participants discontinued from double-blind treatment phase after receiving 240mg loading dose and entered Follow-up phase.) | 3 | 0
Safety Population (Entered From Double-blind Treatment Phase) | 15 | 4 (1 participant who discontinued from double-blind treatment phase after receiving 240mg loading dose and entered Follow-up phase was included under 240mg arm for safety analysis.) | 4 | 0
Entered From Open-label Extension Phase | 438 | 223 | 228 | 0
Safety Population (Entered From Open-label Extension Phase) | 438 | 223 | 228 | 0
Completed | 421 | 217 | 217 | 0
Not Completed | 32 | 11 | 14 | 0
Not completed — Adverse Event | 2 | 0 | 1 | 0
Not completed — Lost to Follow-up | 12 | 5 | 2 | 0
Not completed — Physician Decision | 5 | 1 | 0 | 0
Not completed — Pregnancy | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 12 | 4 | 11 | 0
Period: Israel Addendum
Arm/Group | Placebo | Galcanezumab 120mg | Galcanezumab 240mg | Israel Addendum
Started | 0 (Main study arm.) | 0 (Main study arm.) | 0 (Main study arm.) | 29 (Eligible participants from main study enrolled in Israel addendum.)
Safety Population | 0 | 0 | 0 | 29
Completed | 0 | 0 | 0 | 25
Not Completed | 0 | 0 | 0 | 4
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 4

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Placebo: * Double-blind treatment phase: Participants received placebo once a month by subcutaneous injection for 3 months.
  * Open-label extension phase: After completion of double-blind phase, participants had an option to enter open-label extension phase where they receive 240 mg galcanezumab SC at first month, 120mg at second month followed by 120mg or 240mg once a month (at the discretion of the investigator) for the remaining 7 months.
  * Follow-up phase: After completion or discontinuation from double-blind or open-label extension phases, participants entered follow-up phase where they were observed for 4 months. No treatments administered.
- Total: Total of all reporting groups
Arm/Group | Placebo | Galcanezumab 120mg | Galcanezumab 240mg | Total
Number analyzed (Participants) | 559 | 279 | 279 | 1117
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.61 (12.07) | 39.66 (11.86) | 41.06 (12.36) | 40.98 (12.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 484 | 238 | 228 | 950
  Male | 75 | 41 | 51 | 167
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 122 | 65 | 69 | 256
  Not Hispanic or Latino | 402 | 196 | 194 | 792
  Unknown or Not Reported | 35 | 18 | 16 | 69
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 2 | 0 | 6
  Asian | 26 | 13 | 15 | 54
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 39 | 16 | 17 | 72
  White | 433 | 224 | 225 | 882
  More than one race | 56 | 24 | 21 | 101
  Unknown or Not Reported | 0 | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Argentina | 41 | 20 | 21 | 82
  United States | 314 | 157 | 158 | 629
  Czechia | 25 | 10 | 10 | 45
  United Kingdom | 15 | 7 | 9 | 31
  Spain | 24 | 14 | 12 | 50
  Canada | 8 | 4 | 3 | 15
  Netherlands | 21 | 11 | 11 | 43
  Taiwan | 24 | 12 | 12 | 48
  Italy | 27 | 14 | 15 | 56
  Mexico | 12 | 7 | 5 | 24
  Israel | 20 | 10 | 10 | 40
  Germany | 28 | 13 | 13 | 54
Migraine Headache Days (MHD) [Mean (Standard Deviation); unit: Days per Month] — MHD: A calendar day on which a migraine headache or probable migraine headache occurred. Population: All randomized participants who received at least one dose of study drug.
  Days per Month
    number analyzed (Participants) | 558 | 278 | 277 | 1113
    (all) | 19.55 (4.59) | 19.36 (4.27) | 19.17 (4.60) | 19.41 (4.52)

OUTCOME MEASURES:

1. Primary Outcome: Overall Mean Change From Baseline in the Number of Monthly Migraine Headache Days (MHD)
Description: MHD: A calendar day on which a migraine headache or probable migraine headache occurred.
  Overall mean is derived from the average of months 1 to 3 from mixed model repeated measures (MMRM) model. Least square(LS) Mean was calculated using MMRM model with treatment, pooled country, baseline medication overuse, concurrent prophylaxis use, month, treatment by month, baseline, and baseline by month as fixed effects.
Time Frame: Baseline, Month 1 through Month 3
Population: All randomized participants who received at least one dose of study drug and had baseline and at least one post baseline value.
Measure: Least Squares Mean (Standard Error); unit: Migraine Headache Days per Month
Groups:
- Placebo: Participants received placebo once a month by subcutaneous injection for 3 months.
- Galcanezumab 120mg: Participants received loading dose of 240mg galcanezumab at first dosing visit followed by 120mg of galcanezumab once a month by subcutaneous injection for 2 months.
- Galcanezumab 240mg: Participants received 240 mg of galcanezumab once a month by subcutaneous injection for 3 months.
Arm/Group | Placebo | Galcanezumab 120mg | Galcanezumab 240mg
Number analyzed (Participants) | 538 | 273 | 274
Migraine Headache Days per Month | -2.74 (0.36) | -4.83 (0.44) | -4.62 (0.43)
Statistical Analysis 1: Comparison: Placebo vs Galcanezumab 120mg; Test type: Superiority; p < .001, Mixed Models Analysis; LSMean Difference = -2.09, 95% CI 2-sided [-2.92 to -1.26], Standard Error of Mean 0.42
Statistical Analysis 2: Comparison: Placebo vs Galcanezumab 240mg; Test type: Superiority; p < .001, Mixed Models Analysis; LSMean Difference = -1.88, 95% CI 2-sided [-2.71 to -1.05], Standard Error of Mean 0.42

2. Secondary Outcome: Number of Participants With Reduction From Baseline ≥50%, ≥75% and 100% in Monthly Migraine Headache Days
Description: MHD: A calendar day on which a migraine headache or probable migraine headache occurred.
Time Frame: Baseline, Month 1 through Month 3
Population: All randomized participants who received at least one dose of study drug and had baseline and month 3 measurement.
Measure: Count of Participants; unit: Participants
Groups:
- Galcanezumab 120mg: Participants received loading dose of 240mg of galcanezumab at first dosing visit followed 120mg galcanezumab once a month by subcutaneous injection for 2 months.
Arm/Group | Placebo | Galcanezumab 120mg | Galcanezumab 240mg
Number analyzed (Participants) | 498 | 256 | 262
Participants
  ≥50% | 123 | 90 | 97
  ≥75% | 44 | 34 | 40
  ≥100% | 8 | 4 | 8
Statistical Analysis 1: Comparison: Placebo vs Galcanezumab 120mg; Reduction from Baseline ≥50%,; Test type: Superiority; p = .004, CPRMM; Categorical pseudo likelihood-based repeated measures model (CPRMM); Odds Ratio (OR) = 1.623, 95% CI 2-sided [1.167 to 2.256]
Statistical Analysis 2: Comparison: Placebo vs Galcanezumab 240mg; Reduction from Baseline ≥50%; Test type: Superiority; p < .001, CPRMM; Categorical pseudo likelihood-based repeated measures model (CPRMM); Odds Ratio (OR) = 1.788, 95% CI 2-sided [1.291 to 2.474]
Statistical Analysis 3: Comparison: Placebo vs Galcanezumab 120mg; Reduction from Baseline ≥75%; Test type: Superiority; p = .102, CPRMM; Categorical pseudo likelihood-based repeated measures model (CPRMM); Odds Ratio (OR) = 1.498, 95% CI 2-sided [0.923 to 2.430]
Statistical Analysis 4: Comparison: Placebo vs Galcanezumab 240mg; Reduction from Baseline ≥75%; Test type: Superiority; p = .011, CPRMM; Categorical pseudo likelihood-based repeated measures model (CPRMM); Odds Ratio (OR) = 1.819, 95% CI 2-sided [1.146 to 2.888]
Statistical Analysis 5: Comparison: Placebo vs Galcanezumab 120mg; Reduction from Baseline ≥100%; Test type: Superiority; p = 0.729, CPRMM; Categorical pseudo likelihood-based repeated measures model (CPRMM); Odds Ratio (OR) = 0.761, 95% CI 2-sided [0.163 to 3.563]
Statistical Analysis 6: Comparison: Placebo vs Galcanezumab 240mg; Reduction from Baseline ≥100%; Test type: Superiority; p = .276, CPRMM; Categorical pseudo likelihood-based repeated measures model (CPRMM); Odds Ratio (OR) = 1.897, 95% CI 2-sided [0.600 to 5.998]

3. Secondary Outcome: Mean Change From Baseline in the Migraine-Specific Quality of Life Questionnaire (MSQ) Role-function Restrictive Domain
Description: MSQ v2.1 is a health status instrument, with a 4-week recall period, developed to address physical and emotional limitations of specific concern to individuals with migraine. Addressing the impact of migraine on work or daily activities, relationships with family & friends, leisure time, productivity, concentration, energy, tiredness & feelings. It consists of 14 items that address 3 domains:(1) Role Function-Restrictive (items 1-7);(2) Role Function- Preventive (items 8-11);&(3) Emotional Function (items 12-14).Response options range from "none of the time" (value 1) to "all of the time" (value 6),& are reverse-recoded (value 6 to 1) before the domain scores are calculated. Total raw scores for each domain is the sum of the final item value for all of the items in that domain. After the total raw score is computed for each domain, they are transformed to a 0-100 scale with higher scores indicating a better health status & a positive change in scores reflecting functional improvement.
Time Frame: Baseline, Month 3
Population: All randomized participants who received at least one dose of study drug and had baseline and month 3 measurement.
  LSMean was calculated using MMRM model with treatment, pooled country, baseline medication overuse, concurrent prophylaxis use, month, treatment by month, baseline, and baseline by month as fixed effects.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Galcanezumab 120mg: Participants received loading dose of 240mg galcanezumab at first dosing visit followed 120mg galcanezumab once a month by subcutaneous injection for 2 months.
- Galcanezumab 240mg: Participants received 240mg of galcanezumab once a month by subcutaneous injection for 3 months.
Arm/Group | Placebo | Galcanezumab 120mg | Galcanezumab 240mg
Number analyzed (Participants) | 494 | 252 | 253
units on a scale | 16.76 (1.18) | 21.81 (1.41) | 23.05 (1.63)
Statistical Analysis 1: Comparison: Placebo vs Galcanezumab 120mg; Test type: Superiority; p < .001, Mixed Models Analysis; LSMean Difference = 5.06, 95% CI 2-sided [2.12 to 7.99], Standard Error of Mean 1.50
Statistical Analysis 2: Comparison: Placebo vs Galcanezumab 240mg; Test type: Superiority; p < .001, Mixed Models Analysis; LSMean Difference = 6.29, 95% CI 2-sided [3.03 to 9.55], Standard Error of Mean 1.66

4. Secondary Outcome: Overall Mean Change From Baseline in the Number of Monthly Migraine Headache Days Requiring Medication for the Acute Treatment of Migraine or Headache
Description: Migraine Headache Day (MHD):A calendar day on which a migraine headache or probable migraine headache occurred.
  Overall mean is derived from the average of months 1 to 3 from MMRM model. LSMean was calculated using MMRM model with treatment, pooled country, baseline medication overuse, concurrent prophylaxis use, month, treatment by month,baseline, and baseline by month as fixed effects.
Time Frame: Baseline, Month 1 through Month 3
Population: All randomized participants who received at least one dose of study drug and had baseline and at least one post baseline measurement.
Measure: Least Squares Mean (Standard Error); unit: Days Per Month
Arm/Group | Placebo | Galcanezumab 120mg | Galcanezumab 240mg
Number analyzed (Participants) | 538 | 273 | 274
Days Per Month | -2.23 (0.33) | -4.74 (0.40) | -4.25 (0.40)
Statistical Analysis 1: Comparison: Placebo vs Galcanezumab 120mg; Test type: Superiority; p < .001, Mixed Models Analysis; LSMean Difference = -2.51, 95% CI 2-sided [-3.27 to -1.76], Standard Error of Mean 0.38
Statistical Analysis 2: Comparison: Placebo vs Galcanezumab 240mg; Test type: Superiority; p < .001, Mixed Models Analysis; LSMean Difference = -2.01, 95% CI 2-sided [-2.77 to -1.26], Standard Error of Mean 0.38

5. Secondary Outcome: Mean Change From Baseline in the Patient Global Impression of Severity (PGI-S) Score
Description: PGI-S scale is a participant-rated instrument that measures participants own global impression of their illness severity. The participant was instructed as follows: "Considering migraine as a chronic condition, how would you rate your level of illness?" Response options were from 1 ("normal, not at all ill") to 7 ("extremely ill"). LSMean was calculated using MMRM model with treatment, pooled country, baseline medication overuse, concurrent prophylaxis use, month, treatment by month, baseline, and baseline by month as fixed effects.
Time Frame: Baseline, Month 3
Population: All randomized participants who received at least one dose of study drug and had baseline and month 3 measurement.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Galcanezumab 120mg: Participants received loading dose of 240mg galcanezumab at first dosing visit followed by 120 mg galcanezumab once a month by subcutaneous injection for 2 months.
Arm/Group | Placebo | Galcanezumab 120mg | Galcanezumab 240mg
Number analyzed (Participants) | 494 | 252 | 253
units on a scale | -0.62 (0.08) | -0.76 (0.10) | -0.91 (0.10)
Statistical Analysis 1: Comparison: Placebo vs Galcanezumab 120mg; Test type: Superiority; p = .181, Mixed Models Analysis; LSMean Difference = -0.14, 95% CI 2-sided [-0.34 to 0.06], Standard Error of Mean 0.10
Statistical Analysis 2: Comparison: Placebo vs Galcanezumab 240mg; Test type: Superiority; p = .006, Mixed Models Analysis; LSMean Difference = -0.28, 95% CI 2-sided [-0.48 to -0.08], Standard Error of Mean 0.10

6. Secondary Outcome: Overall Mean Change From Baseline in Headache Hours
Description: Overall mean is derived from the average of months 1 to 3 from MMRM model. LSMean was calculated using MMRM model with treatment, pooled country, baseline medication overuse, concurrent prophylaxis use, month, treatment by month,baseline, and baseline by month as fixed effects.
Time Frame: Baseline, Month 1 through Month 3
Population: All randomized participants who received at least one dose of study drug and had baseline & at least one post baseline measurement.
Measure: Least Squares Mean (Standard Error); unit: Headache Hours per Month
Groups:
- Galcanezumab 120mg: Participants received loading dose of 240 mg galcanezumab at first dosing visit followed 120mg galcanezumab once a month by subcutaneous injection for 2 months.
Arm/Group | Placebo | Galcanezumab 120mg | Galcanezumab 240mg
Number analyzed (Participants) | 538 | 273 | 274
Headache Hours per Month | -13.44 (3.91) | -36.15 (4.74) | -31.53 (4.70)
Statistical Analysis 1: Comparison: Placebo vs Galcanezumab 120mg; Test type: Superiority; p < .001, Mixed Models Analysis; LSMean Difference = -22.71, 95% CI 2-sided [-31.74 to -13.69], Standard Error of Mean 4.60
Statistical Analysis 2: Comparison: Placebo vs Galcanezumab 240mg; Test type: Superiority; p < .001, Mixed Models Analysis; LSMean Difference = -18.09, 95% CI 2-sided [-27.09 to -9.09], Standard Error of Mean 4.58

7. Secondary Outcome: Mean Change From Baseline on the Migraine Disability Assessment Test (MIDAS) Total Score
Description: The MIDAS is a participant-rated scale which was designed to quantify headache-related disability over a 3-month period. This instrument consists of five items that reflect the number of days reported as missing or with reduced productivity at work or home, and the number of days of missed social events. Each item has a numeric response range from 0 to 90 days, if days are missed from work or home they are not counted as days with reduced productivity at work or home. The numeric responses are summed to produce a total score ranging from 0 to 270, in which a higher value is indicative of more disability. LSMean was calculated using Analysis of covariance (ANCOVA) model with last observation carried forward (LOCF) with treatment, pooled country, baseline medication overuse, concurrent prophylaxis use, and baseline value as fixed effects.
Time Frame: Baseline, Month 3
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Galcanezumab 120mg | Galcanezumab 240mg
Number analyzed (Participants) | 504 | 254 | 258
units on a scale | -11.53 (3.38) | -20.27 (4.07) | -17.02 (4.05)
Statistical Analysis 1: Comparison: Placebo vs Galcanezumab 120mg; Test type: Superiority; p = .025, ANCOVA; LSMean Difference = -8.74, 95% CI 2-sided [-16.39 to -1.08], Standard Error of Mean 3.90
Statistical Analysis 2: Comparison: Placebo vs Galcanezumab 240mg; Test type: Superiority; p = .157, ANCOVA; LSMean Difference = -5.49, 95% CI 2-sided [-13.10 to 2.12], Standard Error of Mean 3.88

8. Secondary Outcome: Percentage of Participants Developing Treatment Emergent Anti-drug Antibodies (ADA) to Galcanezumab
Description: A Treatment Emergent Anti-Drug Antibodies (TE ADA) evaluable participant is considered to be TE ADA+ if the participant has at least one post baseline titer that is a 4-fold or greater increase in titer from baseline measurement. If baseline result is ADA Not Present, then the participant is TE ADA+ if there is at least one post baseline result of ADA Present with titer >= 20.
Time Frame: Month 1 through Month 3
Population: All randomized participants who received at least one dose of study drug and had at least one non-missing test result for ADA for each of the baseline period and the post baseline period.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Galcanezumab 120mg | Galcanezumab 240mg
Number analyzed (Participants) | 535 | 264 | 272
Participants | 8 | 7 | 7
Statistical Analysis 1: Comparison: Placebo vs Galcanezumab 120mg; Test type: Superiority; p = .263, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Placebo vs Galcanezumab 240mg; Test type: Superiority; p = .290, Cochran-Mantel-Haenszel

9. Secondary Outcome: Pharmacokinetics (PK): Area Under the Concentration Time Curve (AUC) of Galcanezumab
Description: Pharmacokinetics (PK): Area Under the Concentration Time Curve (AUC) of Galcanezumab.
Time Frame: Baseline through Month 3
Population: Zero participants analyzed. AUC data was not collected as AUC was not pre-specified in protocol.
Arm/Group | Placebo | Galcanezumab 120mg | Galcanezumab 240mg
Number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: Plasma Concentration of Calcitonin Gene-Related Peptide (CGRP)
Description: Plasma Concentration of Calcitonin Gene-Related Peptide (CGRP).
Time Frame: Month 3
Population: All randomized participants who received at least one dose of study drug and had measurable plasma concentrations.
Measure: Mean (Standard Deviation); unit: Nanogram per milliliter (ng/mL)
Groups:
- Galcanezumab 120mg: Participants received loading dose of 240mg galcanezumab at first dosing visit followed by 120mg galcanezumab once a month by subcutaneous injection for 2 months.
Arm/Group | Placebo | Galcanezumab 120mg | Galcanezumab 240mg
Number analyzed (Participants) | 30 | 247 | 253
Nanogram per milliliter (ng/mL) | 0.529 (0.612) | 4.02 (1.70) | 4.85 (1.76)

11. Secondary Outcome: Serum Concentrations of Galcanezumab
Description: Serum concentrations of Galcanezumab
Time Frame: Month 3
Population: All randomized participants who received at least one dose of Galcanezumab and had measurable serum concentrations.
Measure: Mean (Standard Deviation); unit: Nanogram per milliliter (ng/mL)
Groups:
- Galcanezumab 120mg: Participants received loading dose of 240mg galcanezumab at first dosing visit followed 120 mg galcanezumab once a month by subcutaneous injection for 2 months.
Arm/Group | Galcanezumab 120mg | Galcanezumab 240mg
Number analyzed (Participants) | 248 | 254
Nanogram per milliliter (ng/mL) | 16900 (7140) | 29000 (11300)

ADVERSE EVENTS:
Time Frame: Baseline to 16 months for main study plus additional 3 years if enrolled in Israel continued-access addendum.
Description: All participants from safety population. Per protocol, AE analysis was planned per treatment regimen received. Gender specific events only occurring in male or female participants have had the number of participants At Risk adjusted accordingly.
Groups:
- Placebo - Double-Blind Treatment Phase: Participants received placebo once a month by subcutaneous injection for 3 months.
- Galcanezumab 120mg - Double-Blind Treatment Phase: Participants received loading dose of 240mg galcanezumab at first dosing visit followed by 120mg of galcanezumab once a month by subcutaneous injection for 2 months.
- Galcanezumab 240mg - Double-Blind Treatment Phase: Participants received 240 mg of galcanezumab once a month by subcutaneous injection for 3 months.
- Placebo/Galcanezumab - Open-Label Extension Phase: After completion of Placebo double-blind phase, participants had an option to enter open-label extension phase where they received 240 mg galcanezumab SC at first month, 120mg at second month followed by 120mg or 240mg once a month (at the discretion of the investigator) for the remaining 7 months.
- Galcanezumab 120mg/Galcanezumab - Open-Label Extension Phase: After completion of Galcanezumab 120mg double-blind phase, participants had an option to enter open-label extension phase where they received 240mg galcanezumab SC at first month, 120mg at second month followed by 120mg or 240mg once a month (at the discretion of the investigator) for the remaining 7 months.
- Galcanezumab 240mg/Galcanezumab - Open-Label Extension Phase: After completion of Galcanezumab 240mg double-blind phase, participants had an option to enter open-label extension phase where they received 240mg galcanezumab SC at first month, 120mg at second month followed by 120mg or 240mg once a month (at the discretion of the investigator) for the remaining 7 months.
- Placebo - Follow-up Phase: Participants entered follow-up phase from placebo double-blind treatment phase and were observed for 4 months. No treatments administered.
- Galcanezumab 120mg - Follow-up Phase: Participants entered follow-up phase from Galcanezumab 120mg double-blind treatment phase and were observed for 4 months. No treatments administered.
- Galcanezumab 240mg - Follow-up Phase: Participants entered follow-up phase from from Galcanezumab 240mg double-blind treatment phase and were observed for 4 months. No treatments administered.
- Placebo/Galcanezumab - Follow-up Phase: Participants entered follow-up phase from Placebo/Galcanezumabopen-label extension phase and were observed for 4 months. No treatments administered.
- Galcanezumab 120mg/Galcanezumab - Follow-up Phase: Participants entered follow-up phase from Galcanezumab 120mg/Galcanezumab open-label extension phase and were observed for 4 months. No treatments administered.
- Galcanezumab 240mg/Galcanezumab - Follow-up Phase: Participants entered follow-up phase from Galcanezumab 240mg/Galcanezumab open-label extension phase and were observed for 4 months. No treatments administered.
Arm/Group | Placebo - Double-Blind Treatment Phase | Galcanezumab 120mg - Double-Blind Treatment Phase | Galcanezumab 240mg - Double-Blind Treatment Phase | Placebo/Galcanezumab - Open-Label Extension Phase | Galcanezumab 120mg/Galcanezumab - Open-Label Extension Phase | Galcanezumab 240mg/Galcanezumab - Open-Label Extension Phase | Placebo - Follow-up Phase | Galcanezumab 120mg - Follow-up Phase | Galcanezumab 240mg - Follow-up Phase | Placebo/Galcanezumab - Follow-up Phase | Galcanezumab 120mg/Galcanezumab - Follow-up Phase | Galcanezumab 240mg/Galcanezumab - Follow-up Phase | Israel Addendum
All-Cause Mortality (participants affected / at risk) | 0/558 | 0/273 | 0/282 | 0/501 | 0/259 | 0/262 | 0/15 | 0/4 | 0/4 | 0/438 | 0/223 | 0/228 | 0/29
Serious Adverse Events (participants affected / at risk) | 5/558 | 2/273 | 4/282 | 16/501 | 6/259 | 9/262 | 0/15 | 0/4 | 0/4 | 5/438 | 3/223 | 1/228 | 6/29
Other Adverse Events (participants affected / at risk) | 170/558 | 98/273 | 105/282 | 223/501 | 117/259 | 120/262 | 0/15 | 0/4 | 2/4 | 57/438 | 19/223 | 27/228 | 26/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo - Double-Blind Treatment Phase (N=558) | Galcanezumab 120mg - Double-Blind Treatment Phase (N=273) | Galcanezumab 240mg - Double-Blind Treatment Phase (N=282) | Placebo/Galcanezumab - Open-Label Extension Phase (N=501) | Galcanezumab 120mg/Galcanezumab - Open-Label Extension Phase (N=259) | Galcanezumab 240mg/Galcanezumab - Open-Label Extension Phase (N=262) | Placebo - Follow-up Phase (N=15) | Galcanezumab 120mg - Follow-up Phase (N=4) | Galcanezumab 240mg - Follow-up Phase (N=4) | Placebo/Galcanezumab - Follow-up Phase (N=438) | Galcanezumab 120mg/Galcanezumab - Follow-up Phase (N=223) | Galcanezumab 240mg/Galcanezumab - Follow-up Phase (N=228) | Israel Addendum (N=29)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Congenital diaphragmatic hernia (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal adhesions (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alcoholic pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Volvulus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Swelling face (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Complicated appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vestibular neuronitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malignant nipple neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/483 (0) | 0/232 (0) | 0/231 (0) | 0/433 (0) | 0/218 (0) | 0/214 (0) | 0/14 (0) | 0 (0) | 0/3 (0) | 0/376 (0) | 0/186 (0) | 0/184 (0) | 1/25 (1)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Orthostatic intolerance (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1/483 (1) | 0/232 (0) | 0/231 (0) | 0/433 (0) | 0/218 (0) | 0/214 (0) | 0/14 (0) | 0 (0) | 0/3 (0) | 0/376 (0) | 0/186 (0) | 0/184 (0) | 0/25 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Varicose vein (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo - Double-Blind Treatment Phase (N=558) | Galcanezumab 120mg - Double-Blind Treatment Phase (N=273) | Galcanezumab 240mg - Double-Blind Treatment Phase (N=282) | Placebo/Galcanezumab - Open-Label Extension Phase (N=501) | Galcanezumab 120mg/Galcanezumab - Open-Label Extension Phase (N=259) | Galcanezumab 240mg/Galcanezumab - Open-Label Extension Phase (N=262) | Placebo - Follow-up Phase (N=15) | Galcanezumab 120mg - Follow-up Phase (N=4) | Galcanezumab 240mg - Follow-up Phase (N=4) | Placebo/Galcanezumab - Follow-up Phase (N=438) | Galcanezumab 120mg/Galcanezumab - Follow-up Phase (N=223) | Galcanezumab 240mg/Galcanezumab - Follow-up Phase (N=228) | Israel Addendum (N=29)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 2 (2) | 5 (5) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 22 (26) | 9 (12) | 8 (8) | 7 (8) | 4 (5) | 11 (12) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 4 (4)
Asthenia (General disorders) | 0 (0) | 2 (2) | 1 (2) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Fatigue (General disorders) | 6 (6) | 6 (6) | 7 (8) | 7 (7) | 1 (1) | 8 (9) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 4 (4)
Influenza like illness (General disorders) | 3 (3) | 4 (4) | 4 (4) | 5 (5) | 2 (2) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (7)
Injection site erythema (General disorders) | 5 (5) | 4 (5) | 13 (16) | 12 (18) | 6 (6) | 10 (19) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Injection site pain (General disorders) | 24 (32) | 18 (31) | 21 (33) | 8 (10) | 5 (6) | 5 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Injection site reaction (General disorders) | 10 (16) | 8 (13) | 15 (19) | 19 (51) | 21 (56) | 17 (33) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Peripheral swelling (General disorders) | 1 (1) | 1 (1) | 1 (1) | 4 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 1 (1) | 5 (5) | 1 (1) | 5 (5) | 3 (3) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 3 (3) | 5 (5) | 1 (1) | 14 (14) | 7 (7) | 7 (8) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 3 (3) | 3 (3)
Covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Gastroenteritis (Infections and infestations) | 1 (1) | 2 (2) | 2 (2) | 8 (9) | 7 (7) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 2 (2)
Infectious mononucleosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 15 (16) | 0 (0) | 6 (6) | 14 (15) | 17 (21) | 12 (13) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 2 (2) | 4 (4) | 0 (0)
Nasopharyngitis (Infections and infestations) | 24 (26) | 18 (20) | 9 (9) | 45 (55) | 24 (31) | 27 (32) | 0 (0) | 0 (0) | 0 (0) | 11 (11) | 2 (2) | 1 (3) | 5 (6)
Pancreas infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Sinusitis (Infections and infestations) | 5 (5) | 4 (4) | 7 (7) | 16 (17) | 5 (7) | 10 (11) | 0 (0) | 0 (0) | 0 (0) | 7 (7) | 1 (2) | 1 (1) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 14 (14) | 8 (10) | 9 (9) | 27 (31) | 17 (21) | 18 (23) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 2 (2) | 3 (3) | 2 (2)
Urinary tract infection (Infections and infestations) | 6 (6) | 6 (6) | 5 (5) | 29 (33) | 6 (7) | 5 (6) | 0 (0) | 0 (0) | 0 (0) | 9 (10) | 3 (3) | 3 (3) | 4 (4)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (8) | 2 (2) | 5 (5) | 25 (28) | 5 (6) | 7 (9) | 0 (0) | 0 (0) | 0 (0) | 7 (7) | 1 (1) | 0 (0) | 2 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 14 (15) | 8 (9) | 2 (2) | 11 (12) | 13 (13) | 13 (13) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 4 (4) | 0 (0) | 3 (4)
Neck pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 7 (8) | 0 (0) | 3 (3) | 6 (6) | 12 (13) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 1 (1) | 1 (1) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (3) | 2 (2) | 10 (10) | 2 (2) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 3 (3)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 19 (20) | 6 (7) | 9 (10) | 10 (10) | 4 (5) | 7 (11) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (3) | 3 (4)
Headache (Nervous system disorders) | 8 (9) | 4 (4) | 1 (1) | 7 (7) | 5 (5) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (4)
Hypoaesthesia (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Sleep disorder (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Renal cyst (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4) | 4 (4) | 8 (9) | 3 (3) | 9 (9) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 4 (4) | 8 (10) | 5 (5) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 6 (7)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 5 (6) | 4 (4) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4)
Urticaria (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (3) | 0 (0) | 8 (11) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (2) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-01-22): https://cdn.clinicaltrials.gov/large-docs/61/NCT02614261/Prot_000.pdf
  • Statistical Analysis Plan (2017-04-25): https://cdn.clinicaltrials.gov/large-docs/61/NCT02614261/SAP_001.pdf